CLINICAL TRIAL: NCT07262125
Title: Effect of CO2 Pressure on Optic Nerve Sheath Diameter in Laparoscopic Transperitoneal Nephrectomy
Brief Title: Effect of Carbon Dioxide Pressure on Optic Nerve Sheath Diameter in Laparoscopic Transperitoneal Nephrectomy
Acronym: Lap Optic Nerv
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Umut Arslan, MD, Urologist, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Optic Nerve Sheat Laparoscopy
Record Dates: First submitted 2025-09-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Optic Nerve Sheath Diameter; Laparoscopic Nephrectomy
Keywords: optic nerve sheath diameter; laparoscopic nephrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Routine Laparoscopic Pneumoperitoneum (Other): Routine Laparoscopic Pneumoperitoneum of the patients
  Interventions: Diagnostic Test: Optic Nerve Sheath Diameter Measurement

INTERVENTIONS:
Diagnostic Test: Optic Nerve Sheath Diameter Measurement — Optic Nerve Sheath Diameter Measurement, Oxygen saturation and End Tidal CO2 measurements when Pre-operational Supine position, after intubation, Lateral decubitus position, after Pneumoperitoneum, CO2 pressure level at 14-16-18-20 and Post-operational supine position

SUMMARY:
Nephrectomy is a surgical procedure performed for various indications, and with the development and increasing availability of advanced diagnostic techniques, its incidence has been rising. Today, in appropriate cases, laparoscopic surgery is recommended due to its minimally invasive nature and its surgical success rates being comparable to those of open surgery. In laparoscopic surgery, to achieve optimal visualization, a 45° lateral decubitus position is applied, followed by the creation of a pneumoperitoneum using carbon dioxide gas. While the cardiopulmonary effects of this procedure have been shown to be minimal, studies on its intracranial effects are limited. Cerebral perfusion pressure is defined as the difference between mean arterial pressure and either central venous pressure or intracranial pressure, whichever is higher. Intracranial pressure can be assessed non-invasively using ultrasonographic measurement of the Optic Nerve Sheath Diameter (ONSD). The retrobulbar segment of the optic nerve is surrounded by a distensible subarachnoid space, which expands in response to increased intracranial pressure. The effect of increased intra-abdominal pressure during laparoscopic surgery on intracranial pressure, and its impact on ONSD, will be evaluated non-invasively.

In patients scheduled for laparoscopic kidney surgery, the Optic Nerve Sheath Diameter will be measured transorbitally using ultrasonography by the investigator at various stages of the surgery (before anesthesia, after anesthesia, in the lateral decubitus position, during pneumoperitoneum, and at routine intraoperative pressure levels). Additionally, standard monitoring parameters such as pulse rate, blood pressure, oxygen saturation, and End-Tidal CO₂ will be recorded. The Optic Nerve Sheath Diameter, which serves as an indicator of increased intracranial pressure, will be compared with variables such as surgical positioning, BMI, ASA score, and other relevant factors.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 31-69 years.
* Diagnosis of renal cancer (ICD Code C64).
* Planned laparoscopic radical or partial nephrectomy based on current guidelines and patient consent in the Urology Council.

Exclusion Criteria:

* Presence of any condition that prevents transorbital measurement of the optic nerve sheath (e.g., orbital trauma, severe periorbital edema, or ocular abnormalities affecting optic nerve imaging)
* Presence of a medical condition that precludes positioning the patient in a 45-degree lateral decubitus position (e.g., severe scoliosis, respiratory compromise, or spinal instability)
* Known or suspected intracranial pathology that may independently elevate intracranial pressure (e.g., intracranial tumors, hydrocephalus, recent traumatic brain injury)

Ages: 31 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in optic nerve sheath diameter (ONSD) with increasing intraabdominal CO₂ pressure | Preop Supine before intubation → During surgery (baseline supine → lateral decubitus positioning → pneumoperitoneum → each pressure level: 14, 16, 18, 20 mmHg → Postop Supine 5 minutes after extubation of the patient
  Change in optic nerve sheath diameter (ONSD) with increasing intraabdominal CO₂ pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Research and Training Hospital, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atasever AG, Salviz EA, Senturk Ciftci H, Bingul ES, Sivrikoz N, Erdem S, Savran Karadeniz M. The Effects of Lateral 45 degrees Head-Down Position and Carbon Dioxide Pneumoperitoneum on the Optic Nerve Sheath Diameter in Patients Undergoing Laparoscopic Transperitoneal Nephrectomies: A Prospective Observational Study. J Laparoendosc Adv Surg Tech A. 2023 Feb;33(2):171-176. doi: 10.1089/lap.2022.0344. Epub 2022 Aug 25. PMID 36036829
- [Background] Chin JH, Seo H, Lee EH, Lee J, Hong JH, Hwang JH, Kim YK. Sonographic optic nerve sheath diameter as a surrogate measure for intracranial pressure in anesthetized patients in the Trendelenburg position. BMC Anesthesiol. 2015 Mar 31;15:43. doi: 10.1186/s12871-015-0025-9. eCollection 2015. PMID 25861241

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT07262125/Prot_SAP_ICF_000.pdf